CLINICAL TRIAL: NCT07233967
Title: Parent Toolkit to Educate Parents About Pediatric Clinical Research
Brief Title: Parent Resource About Pediatric Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Parentresource-FEA-25-002
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Education
Keywords: Pediatric clinical trials; Parents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Clinical Trials (PCT) Pocket Guide (Experimental): Participants will have access to an intervention between pretest and posttest assessments. The intervention, PCT Pocket Guide, is an online, interactive resource designed to educate parents about pediatric clinical trials and inform their decision-making about their and their child's participation in future pediatric clinical trials.
  Interventions: Behavioral: Pediatric Clinical Trials (PCT) Pocket Guide
- Active Control Resource (Active Comparator): Parents will have access to content from a former NIH-supported website (Children and Clinical Studies) that includes articles and videos about pediatric clinical trials.
  Interventions: Behavioral: Active Control Resource

INTERVENTIONS:
Behavioral: Pediatric Clinical Trials (PCT) Pocket Guide — Parents will interact with a multimedia educational resource that will provide information about pediatric clinical trials, including topics related to participant rights and safety, roles, communication with family, researchers, and healthcare providers, and will provide strategies for shared decision-making.
  Arms: Pediatric Clinical Trials (PCT) Pocket Guide
Behavioral: Active Control Resource — Parents will have access to content from a former NIH-supported website (Children and Clinical Studies) that includes articles and videos about pediatric clinical trials.
  Arms: Active Control Resource

SUMMARY:
The overall aim of this project is to examine the feasibility of a web-based resource for parents to educate them about pediatric clinical research.

DETAILED DESCRIPTION:
Parents (N = 150) of children aged 7-17 years will be recruited from across the United States to participate in a randomized controlled trial. Adult consent will be sought. Participants will be randomized into one of two study arms: intervention and active control. All participants will complete a web-based pretest questionnaire. Participants will then receive access to their randomly assigned resource. Approximately 2-3 weeks after completing the pretest questionnaire, all participants will complete a web-based post-test questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant is a parent or legal guardian of child between ages 7 and 17;
* Participant's child attends school where recruitment flyers have been sent or report that they heard about the study from one of the study recruitment partners;
* Parent has access to a computer or tablet or smart phone with internet connection (as the resource and questionnaires are web-based); and
* Parent is fluent in English or Spanish.

Exclusion Criteria:

* having allowed their child to participate in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knowledge about clinical trials at Week 3 | Baseline and Week 3
  Parents will respond to 8 questions that will assess their factual knowledge about pediatric clinical research (e.g., What does giving 'assent' mean?). Questions are in multiple choice format (some questions have multiple correct answers), and the total score could range from 0-19 correct. Higher scores indicate more knowledge about clinical research.
Change from baseline in attitudes about clinical trials at Week 3 | Baseline and Week 3
  Parents will be asked to respond to 6 questions that assess their positive attitudes about clinical trials (e.g., How do you feel about children and teens participating in clinical trials?; 1=Not good at all; 2=Not very good; 3=Not sure; 4=Good; 5=Very good). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive attitudes toward clinical trials.
Change from baseline in beliefs about clinical trials at Week 3 | Baseline and Week 3
  Parents will be asked to respond to 5 questions about their beliefs about pediatric clinical trials (e.g., I believe that clinical trials are safe for children and teens.; 1=Strongly disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive beliefs about clinical trials.
Change from baseline in likelihood of participation at Week 3 | Baseline and Week 3
  Parents will be asked to respond to one question about the likelihood of allowing their child to participate in a clinical trial (i.e., If your child were asked to be in a clinical trial, how likely would you be to let them participate?; 1 = Not likely; 2 = Somewhat likely; 3 = Moderately likely; 4 = Very likely; 5 = Extremely likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of allowing child to participate in a clinical trial.
Change from baseline in likelihood of fear preventing participation at Week 3 | Baseline and Week 3
  Parents will be asked to respond to one question about the likelihood of their fear preventing them from allowing their child to participate in a clinical trial (i.e., How likely is it that your fearful or anxious feelings could stop you from allowing your child to participate in a clinical trial in the future?; 1 = Not likely; 2 = Somewhat likely; 3 = Moderately likely; 4 = Very likely; 5 = Extremely likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of fear preventing participation in a clinical trial.
Change from baseline in familiarity with clinical trials at Week 3 | Baseline and Week 3
  Parents will be asked to respond to one question about their familiarity with clinical trials [How much do you know about pediatric clinical trials (research studies with children under 18; 1 = I don't know anything about them; 2 = I know a little about them; 3 = I know some things about them; 4 = I know a lot about them; 5 = I know all there is to know about them]. Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater familiarity with pediatric clinical trials.
Change from baseline in willingness to participate at Week 3 | Baseline and Week 3
  Parents will review up to five research protocols related to a fictitious disease ('meditis') and respond to questions about their willingness to let their child participate in each research study (i.e., "If your child had meditis, would you agree to enroll them in this study?"; 1 = Definitely not to 7 = Definitely yes). Responses will be averaged across the five protocols and the minimum scale score is 1 and the maximum scale score is 7. Higher scores indicate greater willingness to allow their child to participate in the research studies.
Change from baseline in decision self-efficacy at Week 3 | Baseline and Week 3
  Parents will be asked to respond to 11 questions about their confidence in obtaining information, asking questions, and making an informed decision about their child's participation in a clinical trial (e.g., Get the facts about the risk and side effects of each choice.; 0 = Not at all confident; 4 = Very confident). Responses will be averaged and the minimum scale score is 0 and the maximum scale score is 4. Higher scores indicate greater decision self-efficacy.
Change from baseline in research trust/mistrust at Week 3 | Baseline and Week 3
  Parents will be asked to respond to 10 questions regarding their trust/mistrust in research (My attitude towards medical research can best be described as positive.; 1 = Strongly disagree; 4 = Strongly agree). The measure has four factors: General Trustworthiness; Perception of Deception; Perception of Exploitation; and Perception of Discriminatory Treatment. Responses will be averaged across each factor and the minimum scale score is 1 and the maximum scale score is 4. Higher scores indicate greater general trustworthiness, greater perceptions of deception, greater perceptions of exploitation, and greater perceptions of discriminatory treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training; Tracy Scull, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No